## Appendix I.9 Statistical Analysis Plan (SAP)

## **Electronic Signature Page**

#### **Full Title**

An open-label extension study to evaluate the long-term safety and tolerability of Lu AE58054 as adjunctive treatment to donepezil in patients with mild-moderate Alzheimer's disease

#### **Short Title**

14861B - Statistical Analysis Plan

Study Number 14861B

The following persons have electronically signed this document

| Server Date and Time | Signed by |
|------------------------------------------|-----------------------|
| 12-Jul-2017 15:00:01 | |
| Reason for Signature | Biostatistic Approval |
| - 10 | |
| 12-Jul-2017 15:11:55 | |
| Reason for Signature | Management Approval |
| 12-Jul-2017 17:28:11 | |
| Reason for Signature | Clinical Approval |
| Reason for Signature | |
| | 1 |
| December Signature | |
| Reason for Signature | |
| Reason for Signature | |
| rtoucon for eignature | |
| Reason for Signature | |
| Reason for Signature | |
| Reason for Signature | |
| Г | |
| D | |
| Reason for Signature | |

Final: Version 1.0 PLUTO ID: CLI 00933680

## Statistical Analysis Plan

# An open-label extension study to evaluate the long-term safety and tolerability of Lu AE58054 as adjunctive treatment to donepezil in patients with mild-moderate Alzheimer's disease

## Idalopirdine (Lu AE58054)

Study No.: 14861B

Sponsor: H. Lundbeck A/S (Lundbeck)

2500 Valby (Copenhagen), Denmark

Biostatistician: Biometrics

SAP date: 10 July 2017

This document is the property of H. Lundbeck A/S and H. Lundbeck A/S is the holder of any and all related intellectual property rights, including, but not limited to, copyrights. This document is confidential. It is not to be copied or distributed to other parties without prior written authorisation from H. Lundbeck A/S.

Trial Site Number: Study Level

Version: 1.0

Pluto ID: CLI\_00933680 Status: Final

LU Study Number: 14861B

## **Table of Contents**

| List | st of Panels | 5 |
|---|---|---|
| List | ist of Abbreviations and Definitions of Terms | 6 |
| 1 | Objectives | <b></b> |
| 2 | Study Design | 8 |
| 3 | Endpoints | 10 |
| 4 | Analysis Sets | 11 |
| 5 | Descriptive Statistics | 11 |
| 6 | Patient Disposition | |
| • | 6.1 Summary of Patient Disposition | |
| | 6.2 Withdrawal | |
| 7 | Demographics and Other Baseline Characteristics | |
| 8 | Recent and Concomitant Medication | |
| 9 | Exposure | |
| 10 | | |
| | 10.1 General Efficacy Analysis Methodology | |
| | 10.2 Exploratory Analysis of Efficacy | |
| 11 | $oldsymbol{arepsilon}$ | |
| | 11.1 Adverse Events | |
| | 11.1.1 General Methodology for Adverse Events | |
| | 11.1.2 Coding of Adverse Events | |
| | 11.1.3 Classification of Adverse Events | |
| | 11.1.4 Allocation of TEAEs to Treatment Periods | |
| | 11.1.5 All Adverse Events | |
| | 11.1.6 Treatment-emergent Adverse Events | |
| | 11.1.7 Deaths | |
| | 11.1.8 Serious Adverse Events | |
| | 11.1.9 Adverse Events Leading to Withdrawal | |
| | 11.1.10 Adverse Events Leading to Dose Reduction of IMP | |
| | 11.1.11 Adverse Events of Special Interest | |
| | 11.2 General Methodology for Other Safety Data | |
| | 11.3 Clinical Safety Laboratory Test Data | |
| | 11.3.1 Data Presentation | |
| | 11.3.2 Urinalysis | |
| | 11.3.3 Evaluation of Potential Drug-induced Liver Injury (DILI | |
| | 11.4 Vital Signs and Weight | |
| | 11.5 ECGs | |
| | 11.6 Columbia-Suicide Severity Rating Scale (C-SSRS) | 22 |

Trial Site Number: Study Level


| 12 | Phar | macokinetic/Pharmacodynamic Analyses | 23 |
|---|---|---|---|
| 13 | Heal | th Economic Analyses | 23 |
| 14 | | im Analyses | |
| 15 | | ple Size Considerations | |
| 16 | Data | and Analysis Standards and Statistical Software | <b>2</b> 4 |
| 17 | Chai | nges to Analyses Specified in the Protocol | <b>2</b> 4 |
| 18 | Deta | ils on Data Handling | 24 |
| | | Definition of Baseline | |
| | 18.2 | Derived Variables | 25 |
| | | 18.2.1 MMSE Total Score and MMSE Stratum | 25 |
| | | 18.2.2 ADAS-Cog Total Score | |
| | | 18.2.3 ADCS-ADL <sub>23</sub> Total Score | |
| | | 18.2.4 NPI Total Score and Individual Items | |
| | 18.3 | Assigning Data to Visits | |
| | | 18.3.1 Rating Scales | |
| | | 18.3.2 Safety Variables | |
| | 18.4 | Handling of Missing or Incomplete Dates/Times | |
| | | 18.4.1 IMP Start and Stop Dates | |
| | | 18.4.2 Withdrawal Date | |
| | | 18.4.3 Medical Disorder Start and Stop Dates | |
| | | 18.4.4 Adverse Event Start and Stop Dates | |
| | 18.5 | | |
| Refe | erences | | 35 |


## Appendices

| Appendix I | Statistical Analysis Plan Authentication and Authorisation | 30 |
|---|---|---|
| Appendix II | Study Flow Chart | 38 |
| Appendix III | SAS® Code | 4 |
| Appendix IV | PCS Criteria | 40 |

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final

## **List of Panels**

| Panel 1 | Study Design: Open-label treatment period | 9 |
|---|---|---|
| Panel 2 | Study Design: Open-label treatment period with memantine | 10 |
| Panel 3 | Graphical Presentations for the Liver Function Tests | 19 |
| Panel 4 | Graphical Presentations for Vital Signs and Weight | 2 |
| Panel 5 | Graphical Presentations for ECG Parameters | 22 |
| Panel 6 | C-SSRS Scores | 23 |
| Panel 7 | Definition of ADAS-Cog Item Scores | 26 |
| Panel 8 | ADCS-ADL <sub>23</sub> Items | 28 |
| Panel 9 | Visit Windows for Efficacy Assessments (open-label treatment period) | 32 |
| Panel 10 | Visit Windows for MMSE | 32 |
| Panel 11 | Visit Windows for Safety Assessments | 33 |

#### List of Abbreviations and Definitions of Terms

γGT γ-glutamyl transferase AD Alzheimer's disease

ADAS-Cog Alzheimer's Disease Assessment Scale, cognitive subscale

ADCS-ADL<sub>23</sub> Alzheimer's Disease Cooperative Study – Activities of Daily Living Inventory
ADCS-CGIC Alzheimer's Disease Cooperative Study – Clinical Global Impression of Change

ADL Activities of Daily Living

AE adverse event

ALT alanine aminotransferase
ALP alkaline phosphatase
APTS all-patients-treated set
AST aspartate aminotransferase
ATC anatomical therapeutic chemical

BMI body mass index
BP blood pressure
BUN blood urea nitrogen

CRA clinical research associate

CRF case report form CRP C-reactive protein

C-SSRS Columbia-Suicide Severity Rating Scale

ECG electrocardiogram

eCRF electronic case report form

FDA United States Food and Drug Administration

IMP investigational medicinal product

INR international normalised ratio of prothrombin time

MMRM mixed model for repeated measurements

MMSE Mini Mental State Examination
NPI Neuropsychiatric Inventory

PBO placebo

PCS potentially clinically significant

PR specific ECG interval describing atrioventricular conduction

QP qualified person

QRS specific ECG interval describing ventricular depolarisation

QTcF heart-rate corrected QT interval using Fridericia's correction formula

REML restricted maximum likelihood

RUD Lite Resource Utilisation in Dementia Lite SADs Lundbeck Standard Analysis Datasets

SAE serious adverse event

SDTM Standard Data Tabulation Model


LU Study Number: 14861B Pluto ID: CLI 00933680

Status: Final


Trial Site Number: Study Level

SOC system organ class

TEAE treatment-emergent adverse event

ULN upper limit of normal

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final Version: 1.0

Trial Site Number: Study Level

## 1 Objectives

#### 1.1 Primary Objective

Open-label treatment period:

To evaluate the long term safety and tolerability of idalopirdine as adjunctive therapy to donepezil in patients with mild-moderate AD.

*Open-label treatment period with memantine (sub-study):* 

To evaluate the safety and tolerability of concomitant treatment with idalopirdine, memantine and donepezil in patients with mild-moderate AD.

#### 1.2 Secondary Objective

Open-label treatment period:

To evaluate the long-term disease development during treatment with idalopirdine as adjunctive therapy to donepezil in patients with mild-moderate AD.

*Open-label treatment period with memantine (sub-study):* 

To evaluate the disease development during concomitant treatment with idalopirdine, memantine and donepezil in patients with mild-moderate AD.

#### 1.3 Other Objectives

Open-label treatment period with memantine (sub-study):

To explore population pharmacokinetics.

## 2 Study Design

This is an interventional, multi-national, multi-site, open-label extension study in patients with mild to moderate AD who completed the 24-week "lead-in" double-blind, placebo controlled clinical studies 14861A and 14862A (from now on these studies will be referred to as "lead-in study" in the document). Randomized, blinded treatment in lead-in study will remain blinded to sites, CRAs, patients, and investigators until patients have completed the extension study (the sponsor will generally be un-blinded after unblinding of 14861A and 14862A occurs).

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Patients completing the open-label treatment period and who will not continue into the 24-week open-label memantine sub-study (described below) will enter a 4-week safety follow-up period. Thus the total study duration of the open-label treatment period per patient from Baseline II (Visit 1 of the open-label treatment period and Visit 7 of the lead-in study) to the end of the follow-up will be approximately 32 weeks.

Some sites will be participating in the open-label treatment period with memantine (substudy). In total, 100 patients who have completed the open-label treatment period will be recruited for the for the memantine sub-study. For these patients, the study will include two consecutive periods:

- Open-label treatment period (initial 28-week period): 28-weeks with idalopirdine 60 mg/day as adjunctive treatment to donepezil (10 mg/day). The dose of idalopirdine can be decreased to 30 mg/day if 60 mg/day is not well tolerated in the opinion of the investigator. The Baseline Visit of this period (Baseline II) will be the same visit as Visit 7 (Completion Visit) in the lead-in studies.
- Open-label treatment period with memantine (sub-study): 24-weeks with idalopirdine 60 mg/day (or 30 mg/day) [continuation of dose used in open-label treatment period] as adjunctive treatment to donepezil hydrochloride 10 mg/day and memantine (patient's individualised maintenance dose, including a titration phase of up to 3 weeks). Memantine should be prescribed according to investigator's judgement and the initial dose may be changed at any time throughout the course of the study, if clinically indicated in the opinion of the investigator. The Baseline Visit of this period (Baseline III) will be the same visit as Visit 6 in the open-label treatment period.

Patients completing the two consecutive treatment periods will enter a 4-week safety follow-up period. Thus the total study duration per patient in the sub-study from Baseline II to the end of the follow-up will be approximately 56 weeks.

The study design is presented in Panel 1 and Panel 2 and the scheduled assessments are summarised in Appendix II.



Trial Site Number: Study Level

Panel 1 Study Design: Open-label treatment period

LU Study Number: 14861B Pluto ID: CLI\_00933680



Panel 2 Study Design: Open-label treatment period with memantine

## 3 Endpoints

Secondary efficacy enpoints in the open label treatment period

- Change from Baseline I to week 52 (extension week 28) in Alzheimer's disease Assessment Scale-cognitive subscale (ADAS-cog) total score
- Change from Baseline II to week 52 (extension week 28) in ADAS-cog total score
- Alzheimer's disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC) at week 52 (extension week 28)
- Change from Baseline I to week 52 in Change from baseline to Week 24 (extension week 28) in Alzheimer's disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL<sub>23</sub>) total score
- Change from Baseline II to week 52 (extension week 28) in ADCS-ADL<sub>23</sub> total score
- Change from Baseline I to week 52 (extension week 28) in Neuropsychiatric Inventory (NPI) total score and NPI single items
- Change from Baseline II to week 52 (extension week 28) in NPI total score and NPI single items
- Change from Baseline I to week 52 (extension week 28) in Mini Mental State Examination (MMSE) total score
- Change from Baseline II to week 52 (extension week 28) in MMSE total score

Secondary efficacy enpoint in the open label treatment period with memantine

• Change from Baseline III to week 24 in MMSE total score

Safety endpoints

• Adverse events (AEs)

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

- Clinical safety laboratory tests
- Vital signs
- Weight
- Electrocardiograms (ECGs)
- Columbia Suicide Severity Rating Scale (C-SSRS)

#### Other endpoints

• Plasma concentrations of idalopirdine and memantine in the open label treatment period with memantine

## 4 Analysis Sets

The following analysis set will be used to analyse and present data:

The sets of patients to be analysed are defined as follows:

Open label treatment period

- all-patients-enrolled set (APES) all patients enrolled in the open-label treatment period
- *all-patients-treated set* (APTS) all patients in APES who took at least one dose of IMP in the open-label treatment period

Open label treatment period with memantine

- *all-patients-enrolled set 2* (APES2) all patients who enrolled in the open-label treatment period with memantine
- *all-patients-treated set 2* (APTS2) all patients in APES2 who took at least one dose of IMP or memantine in the open-label treatment period with memantine.

Each patient will be classified according to these definitions based on information in data, and no Classification Meeting will be held.

If not otherwise specified, tables, figures, and listings will be based on the APTS for the open-label treatment period, and on APTS2 for the open-label treatment period with memantine.

## 5 Descriptive Statistics

Unless otherwise specified, summary statistics (n, arithmetic mean, standard deviation [SD], median, lower and upper quartiles, minimum and maximum values) will be presented for continuous variables, and counts and, if relevant, percentages will be presented for categorical variables.

Tables and figures for the open label treatment period will be presented by lead-in treatment group and in total.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Unless otherwise specified, data listings will include lead-in treatment group (placebo or idalopirdine [dose 10mg, 30mg, or 60mg]), site, patient screening number (from lead-in study), and lead-in study-Baseline I information on sex, age, race, and weight.

## **6** Patient Disposition

#### 6.1 Summary of Patient Disposition

Patient disposition in the open label-treatment period will be summarised by lead-in study and in total, and include the number of patients in each analysis set defined for the period, and the number of patients in the APTS who completed or withdrew from treatment. The corresponding summary will be generated for the open-label treatment period with memantine for the total study.

#### 6.2 Withdrawal

The number of patients who withdrew from the open-label treatment period will be summarised by primary reason for withdrawal as well as by all reasons for withdrawal.. Similar summaries will be created for the open-label treatment period with memantine. The summaries will also be presented by lead-in study for the open-label treatment period.

Patients who withdrew from treatment during the open-label treatment period will be listed and the listing will include the number of days on idalopirdine in the open-label treatment period, the primary reason for withdrawal from treatment, and all reasons for withdrawal from treatment. A similar listing will be created for patients who withdrew from treatment during the open-label treatment period with memantine.

## 7 Demographics and Other Baseline Characteristics

Demographics and baseline characteristics at Baseline I will be summarised for patients in the APTS and the APTS2.

Demographics (sex, age, ethnicity, and race), patient characteristics (weight, height, BMI), and efficacy variables at Baseline I will be summarised.

Past and concurrent medical, neurological, and psychiatric disorders at the lead-in study Screening Visit (coded using the Medical Dictionary for Regulatory Activities [MedDRA], Version 19.0 or later), will be summarised.

The summaries will also be presented by lead-in study for the APTS.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

#### 8 Recent and Concomitant Medication

Recent and concomitant medication will be coded using the WHO Drug Dictionary (WHO-DDE), version WHO ATC MAR16., and summarised by anatomical therapeutic chemical (ATC) code, and generic drug name.

For the open label treatment period summaries will be prepared for:

- Concomitant medication continued after Baseline II
- concomitant medication started after Baseline II and at or before Baseline III for patients in APES2

For the open label treatment period with memantine summaries will be prepared for;

- concomitant medication continued after Baseline III
- concomitant medication started after Baseline III

A listing will be created that includes information about memantine dosages over the course of the open label treatment period with memantine.

## 9 Exposure

Exposure to IMP in this study will be defined as: date of last dose of IMP – date of first dose of IMP + 1

For details about handling of missing IMP start or stop date, see section 18.4.1 (IMP start and stop date)

Exposure to IMP in each treatment period will be summarised using descriptive statistics, and include the patient years of exposure (PYE). PYE will be calculated as the sum of the number of days of exposure to IMP for each patient, divided by 365.25 days.

In addition, exposure to IMP in each treatment period will be categorised into day intervals. The intervals for the open-label treatment period are the following:  $(1-28\ [0-1\ month], 29-56\ [1-2\ months], 57-84\ [2-3\ months], 85-126\ [3-4.5\ months], 127-168\ [4.5-6\ months], 169-252\ [6-9\ months].$  The intervals for the open-label treatment period with memantine are the following:  $(1-168\ [0-6\ months], 169-252\ [6-9\ months], 253-364\ [9-12\ months], 365-448\ [12-15\ months])$ . Missing values of exposure will not be imputed.

Number and percentage of patients with dose reduction of IMP to 30 mg/day in the open-label treatment period will be summarised. The mean dose of IMP will be calculated for each patient and summarised (mean, median, and lower and upper quartiles). Categorical summaries of patients' dosage at each visit will be presented as well.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

## 10 Efficacy

#### 10.1 General Efficacy Analysis Methodology

All analyses will be performed by lead-in study.

For the open label treatment period, absolute scores, change from Baseline I scores, and change from Baseline II scores for the efficacy variables will be summarised by visit week. The summaries of absolute scores and change from Baseline I scores will include data from the lead-in study and the open-label treatment period.

For the open label treatment period with memantine, absolute score and change from Baseline Baseline III in MMSE total score will be summarised by visit week.

All the p-values will be based on two-sided tests; the confidence intervals (CIs) will be two-sided.

Nominal p-values will be presented together with nominal 95% CIs.

#### 10.2 Exploratory Analysis of Efficacy

Changes from baseline I in ADAS-Cog total score, ADCS-ADL<sub>23</sub> total score, NPI total score, NPI individual items, and MMSE total score will be analysed using a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM) approach. Baseline will be defined as the baseline in the lead-in study (Baseline I). The model will include data from visits in both the lead-in study and the open label treatment period. The model will include the fixed categorical effects of treatment group in the lead-in study, country, visit week, treatment-by-week interaction, MMSE-stratum ( $<19, \ge19$ ) at baseline I, and MMSE-stratum at baseline I-by-visit interaction and the continuous covariates of baseline score and baseline score-by-visit interaction.

In all analyses, an unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis will be based on the missing-at-random (MAR) assumption and performed using all available observations (observed cases [OC] data).

Line plots will be created to illustrate the MMRM estimates of least squares means by visit week. ADCS-CGIC will be analysed using the same methodology, using the scores at each visit and the ADCS-CGIC score at Baseline I in the lead-in study as baseline.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

## 11 Safety

#### 11.1 Adverse Events

#### 11.1.1 General Methodology for Adverse Events

The tables for the open label treatment periodwill be sorted in descending order by the percentage of patients in the lead-in IDL 60 mg group. Unless otherwise specified, the summaries of adverse events will include the total number and percentage of patients with an adverse event. For sex-specific preferred terms, the denominator in the % calculations will be the number of patients of that sex. Sex-specific preferred terms will be marked in the summaries.

In summaries of adverse events presented by intensity, the maximum intensity of the adverse event in the treatment period will be used for patients who have more than one intensity of that event. Adverse events for which information on intensity is missing will be classified as *severe*.

Listings of adverse events will be sorted by lead-in study treatment group, site, patient screening number (from lead-in study), and adverse event start date and include preferred term, investigator term, adverse event start date, days since first dose of IMP in the treatment period, duration of the adverse event in the treatment period, date of death, action taken, causality, intensity, seriousness, and outcome. For adverse events that change in intensity, each intensity will be included.

#### 11.1.2 Coding of Adverse Events

Adverse events will be coded using MedDRA, Version 19.0, or later.

#### 11.1.3 Classification of Adverse Events

Adverse events will be classified according to the time of onset of the adverse event: treatment-emergent adverse event (TEAE) – an adverse event that starts or increases in intensity after the date of Baseline II.

An adverse event is considered causally related to the use of the IMP when the causality assessment by the investigator is *probable* or *possible*.

#### 11.1.4 Allocation of TEAEs to Treatment Periods

TEAEs will be allocated to treatment periods according to the time of onset of the adverse event:

• *adverse event in the open-label treatment period* – an adverse event that starts or increases in intensity after the date of Baseline II and at or before the date of the last protocol-

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

- specified contact in the study for patients not continuing into the open-label treatment period with memantine, and at or before the date of Baseline III for patients in the APES2.
- adverse event in the open-label treatment period with memantine an adverse event that starts or increases in intensity after the date of Baseline III and at or before the date of the last protocol-specified contact in the study.

Note, the completion Visit in the lead-in studies are the same as the Baseline II Visit in the extension study, and adverse events ongoing or starting at Baseline II and not increasing intensity will only be reported in the lead-in study.

All tables and listings will be presented separately for adverse events in the open label treatment period, and the open label treatment period with memantine.

#### 11.1.5 All Adverse Events

All adverse events will be listed for the APES and APES2.

An overview of the PYE, numbers, and percentages of patients with TEAEs, serious adverse events (SAEs), adverse events leading to withdrawal, or patients who died will be provided. For TEAEs, SAEs, and adverse events leading to withdrawal, the total number of events will be included.

#### 11.1.6 Treatment-emergent Adverse Events

The following summaries will be provided:

- TEAEs by SOC and preferred term (only for open label treatment period)
- TEAEs by preferred term
- TEAEs with an incidence >3% by preferred term
- causally related TEAEs by SOC and preferred term TEAEs by intensity (*mild/moderate/severe*) and preferred term
- causally related TEAEs by intensity and preferred term (only for open label treatment period)

#### 11.1.7 **Deaths**

All adverse events for patients who died will be listed.

#### 11.1.8 Serious Adverse Events

All SAEs will be listed.

Treatment-emergent SAEs will be summarised by preferred term. For the open label treatment period the summary will also be generated by SOC and preferred term.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

#### 11.1.9 Adverse Events Leading to Withdrawal

All adverse events leading to withdrawal will be listed.

TEAEs leading to withdrawal will be summarised by preferred term. For the open label treatment period the summary will also be generated by SOC and preferred term.

#### 11.1.10 Adverse Events Leading to Dose Reduction of IMP

Adverse events leading to dose reduction of idalopirdine in the open label treatment period will be listed.

Adverse events leading to dose reduction of idalopirdine in the open label treatment period will be summarised by preferred term.

#### 11.1.11 Adverse Events of Special Interest

The following standardized MedDRA queries (SMQ) will be summarised in total and by preferred term:

- Convulsions (narrow scope)
- Drug-related hepatic disorders -comprehensive search
- Haemorrhages (broad scope)

#### 11.2 General Methodology for Other Safety Data

The denominators for the summaries of a given variable will be based on the number of patients with non-missing values at a given visit or during the assessment period.

Descriptive statistics for the safety variables in the open label treatment period, absolute values changes from both Baseline I and Baseline II, will be presented by visit and the last post-baseline assessment in the treatment period.

For the open-label treatment period with memantine, summaries will be presented for absolute values and change from Baseline III by visit and last assessment in the treatment period.

The number and percentage of patients with at least one PCS value at any post-Baseline II assessment in the open-label treatment period will be summarised by variable. The number and percentage of patients with at least one PCS value at any post-Baseline III assessment in the open-label treatment period with memantine will be summarised by variable . All available assessments will be included in the evaluation of PCS values (scheduled, reassessments, and unscheduled). For tests where PCS is defined as a change, the summaries will be prepared both for PCS compared to baseline I and baseline II for the open label treatment period.

For patients with post-baseline II PCS values (compared to baseline II) in the open-label treatment period, listings will be provided including all available values for the variable, with

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680


flagging of PCS values and out-of-reference-range values. The corresponding listings will be prepared for the open label treatment period with memantine.

All adverse events for patients with post-baseline II PCS value (compared to baseline II) in the open-label treatment periods will be listed by lead-in treatment group and patient screening number and include the PCS value; investigator term and preferred term for the adverse event; and intensity, seriousness, causality, action taken, outcome, start date, and duration of the adverse event; and days since first dose of IMP at the time of onset of the adverse event. The PCS value will be listed next to any adverse events occurring in the same visit window; the PCS values and adverse events will be listed in chronological order according to assessment date and the start date of the adverse event. The corresponding listings will be presented for the open-label treatment period with memantine.

#### 11.3 Clinical Safety Laboratory Test Data

#### 11.3.1 Data Presentation

The PCS criteria for the clinical safety laboratory tests are in Table 1.

All the clinical safety laboratory test values will be presented in conventional and/or Système International (SI) units.

The summary statistics for GGT, ALT, AST, ALP, Bilirubin, and eosinophils will be presented in a separate tables, including worst (highest) post-Baseline II assessment during the open-label treatment period or post-Baseline III assessment during the open-label treatment period with memantine. All available assessments will be included in the evaluation of the worst assessment.

Graphical presentations of gamma glutamyl transferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and bilirubin (BILI) are described Panel 3 (further graphical presentations of ALT, AST, ALP, and BILI will be done in the evaluation of drug-induced liver injury).

LU Study Number: 14861B Pluto ID: CLI 00933680

Status: Final

Trial Site Number: Study Level


**Panel 3** Graphical Presentations for the Liver Function Tests

| <b>Laboratory Test</b> | Measure | Patient Selection | Line Plot |
|---|---|---|---|
| Open-label treatm | Open-label treatment period | | |
| GGT | Absolute measure | Patients with a post-Baseline II value of GGT ≥200 | $\sqrt{}$ |
| ALT | Absolute measure | Patients with a post-Baseline II value out of upper reference range for ALT | $\sqrt{}$ |
| AST | Absolute measure | Patients with a post-Baseline II value out of upper reference range for AST | $\sqrt{}$ |
| ALP | Absolute measure | Patients with a post-Baseline II value out of upper reference range for ALP | $\sqrt{}$ |
| BILI | Absolute measure | Patients with a post-Baseline II value out of upper reference range for BILI | $\sqrt{}$ |
| Open-label treatm | ent period with men | nantine | |
| GGT | Absolute measure | Patients with a post-Baseline III value of GGT≥200 | $\sqrt{}$ |
| ALT | Absolute measure | Patients with a post-Baseline III value out of upper reference range for ALT | $\sqrt{}$ |
| AST | Absolute measure | Patients with a post-Baseline III value out of upper reference range for AST | $\sqrt{}$ |
| ALP | Absolute measure | Patients with a post-Baseline III value out of upper reference range for AP | $\sqrt{}$ |
| BILI | Absolute measure | Patients with a post-Baseline III value out of upper reference range for BILI | $\sqrt{}$ |

#### 11.3.2 Urinalysis

For tests based on urine dipsticks, the results are categorical, and the number and percentage of patients will be summarised for each test by visit week and last assessment in each treatment period.

#### 11.3.3 Evaluation of Potential Drug-induced Liver Injury (DILI)

Signals of DILI post-Baseline II for the open label treatment period and post Baseline III for the open label treatment period with memantine will be assessed according to the FDA guideline<sup>1</sup>, as well as by using additional criteria, as described below:

The number and percentage of patients post-Baseline II/Baseline III in the categories below for AST/ALT, and AST and ALT separately will be summarised:


- ULN < value  $\le 1.5$ xULN
- $1.5xULN < value \le 2xULN$
- $2xULN < value \le 3xULN$
- $3xULN < value \le 5xULN$
- $5xULN < value \le 10xULN$
- $10xULN < value \le 20xULN$

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Status: Final

#### • 20xULN < value

The number and percentage of patients post-Baseline II/Baseline III in the categories below for ALP and Bilirubin will be summarised:

- ULN<value ≤1.5xULN
- 1.5xULN< value <2xULN
- 2xULN< value ≤3xULN
- value >3xULN

In the summaries, each patient should be counted only once using the worst post-Baseline II/Baseline III assessment.

The cumulative number and percentage of patients post-baseline in the categories will also be summarised for each treatment period.

Number and percentage of patients fulfilling the joint criteria below post-baseline II/Baseline III will be summarised:

- (PEAK AST OR PEAK ALT>3xULN ) AND PEAK BILI>2xULN AND PEAK ALP>1.5xULN
- (PEAK AST OR PEAK ALT>3xULN ) AND PEAK BILI>2xULN AND PEAK ALP<1.5xULN
- PEAK GGT>200 (IU/L) without (PEAK AST OR PEAK ALT OR PEAK ALP>2xULN)
- Number and percentage of patients with a post-Baseline II /Baseline III value ≥5% for Beosinophils/leukocytes (ESOLE) will be summarised.

Evaluation of potential Drug-Induced Serious Hepatotoxicity (eDISH) will also be done by plots. Scatter plots of peak ALT/AST versus peak BILI in the treatment period (note that this means that the peak ALT/AST and the peak BILI may not occur at the same assessment timepoint). The values will be normalised by the ULN (unit xULN) and the X and Y-axes will be on log scale. The plot will include a reference line for ALT/AST values >3xULN, and a reference line for BILI values>2xULN. Four quadrants are defined by the reference lines, where the right upper quadrant being the most specific indicator for a drug's potential for causing serious liver injury (Hy's law quadrant). The plot will include number of patients in each quadrant.

Subject line plots with values-by-time for ALT, AST, ALP, Bilirubin, eosinophils, and GGT (overlaid in the same plot) will be generated for patients with ALT/AST > 1xULN post-baseline II/Baseline III. The test values will be normalised by the ULN (unit xULN) and the Y-axis will be on log scale. The time will be days since Baseline II/Baseline III, and reference lines for the day of first-and last IMP intake in the treatment period will be included. All assessments will be included. If there is more than one assessment at the same time point for a test, the maximum value will be used. A corresponding plot will be generated for patients with ALT/AST > 3xULN post-baseline I in the lead-in study or the open-label treatment period, where values in the lead-in treatment period and the open-label treatment will be included.


LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Status: Final


Conditional correlations of values adjusted for patient average level (mean value for each patient within each treatment period subtracted from the subject values at each visit within the treatment period) of ALT, AST, ALP, and bilirubin versus eosinophils will be generated as tables and scatter plots for:

- All patients
- Patients with a post-baseline II/Baseline III value of ALT/AST>2xULN
- Patients with a post-baseline II/Baseline IIIvalue of ALT/AST>3xULN

Patients in the APTS with a post-Baseline II/Baseline III value of GGT, ALT, AST, ALP, bilirubin, >1xULN will be listed, and the listing will include all available ALT, AST, BILI, ALP, GGT, and EOSLE values, sorted by completion/withdrawal status, treatment group, site, subject number, assessment date and time.

#### 11.4 Vital Signs and Weight

The PCS criteria for vital signs and weight are in Table 2.

An overview of the graphical presentations is provided in Panel 4.

Panel 4 Graphical Presentations for Vital Signs and Weight

| Variable | Measure | Patient Selection | Line Plot |
|---|---|---|---|
| Weight | Absolute value | Patients with a post-Baseline II PCS Low Value<br>Compared to Baseline I in the open label<br>treatment period | V |
| Weight | Absolute value | Patients with a post-baseline II PCS Low Value<br>Compared to Baseline II in the Open-label<br>Treatment Period | $\sqrt{}$ |
| Weight | Absolute value | Patients with a post-baseline III PCS Low Value Compared to Baseline I | $\sqrt{}$ |
| Weight | Absolute value | Patients with a post-baseline III PCS Low Value Compared to Baseline III | $\sqrt{}$ |

#### 11.5 ECGs

The PCS criteria for the ECG parameters are in Table 3.

An overview of the graphical presentations for the ECG parameters is provided in Panel 5.

LU Study Number: 14861B Pluto ID: CLI 00933680

Status: Final

Trial Site Number: Study Level


That Site Number. Study Level

**Panel 5** Graphical Presentations for ECG Parameters

| Parameter | Measure | Patient Selection | Line Plot |
|---|---|---|---|
| Heart ate | Absolute value | Patients with a post-Baseline II PCS value compared to Baseline I in the open label treatment period | V |
| Heart ate | Absolute value | Patients with a post-Baseline II PCS value compared to Baseline II in the open label treatment period | $\sqrt{}$ |
| QTcF | Absolute value | Patients with a post-Baseline II PCS value compared to Baseline I in the open label treatment period | $\sqrt{}$ |
| QTcF | Absolute value | Patients with a post-Baseline II PCS value compared to Baseline II in the open label treatment period | $\checkmark$ |
| Heart rate | Absolute value | Patients with a post-Baseline III PCS value compared to Baseline I | $\sqrt{}$ |
| Heart rate | Absolute value | Patients with a post-Baseline III PCS value compared to Baseline III | $\sqrt{}$ |
| QTcF | Absolute value | Patients with a post-Baseline III PCS value compared to Baseline I | $\sqrt{}$ |
| QTcF | Absolute value | Patients with a post-Baseline III PCS value compared to Baseline III | $\checkmark$ |

#### 11.6 Columbia-Suicide Severity Rating Scale (C-SSRS)

For all visits, the C-SSRS was assessed using the Since Last Visit Version that collects information for a pre-specified, limited period.

The C-SSRS scores will be summarised (as described below) for open-label treatment period and open label treatment period with memantine for patients with at least one post-Baseline II/Baseline III, regardless of whether they had a Baseline II/Baseline III assessment.

Missing C-SSRS scores will not be imputed.

The C-SSRS items are described in Panel 6. Patients with *no suicidal ideation or behaviour* are those who answered "No" to all items for *suicidal ideation* and *suicidal behaviour*. For each evaluation (baseline II and post-baseline II for the open label treatment period, and baseline III, and post-baseline III for the open-label treatment period with memantine), the most severe event per patient related to *suicidal ideation* and *suicidial behaviour* will be summarised.

In the C-SSRS, *non-suicidal self-injurious* behaviour is captured as a different behaviour, and regarded independently of reported *suicidal ideation* and *suicidal behaviour* events. Positive responses to *non-suicidal self-injurious behaviour* will be summarised.

LU Study Number: 14861B Pluto ID: CLI 00933680

Status: Final

Trial Site Number: Study Level


| Panel 6 | C-SSRS Scores |
|-----------|-----------------|
| I AIICI O | ( -00110 0001 C |

| aCRF Item | Description |
|---|---|
| | Suicidal Ideation |
| CSSRS01 | Wish to be dead |
| CSSRS02 | Non-specific active suicidal thoughts |
| CSSRS03 | Active suicidal ideation with any methods (not plan) without intent to act |
| CSSRS04 | Active suicidal ideation with some intent to act, without specific plan |
| CSSRS05 | Active suicidal ideation with specific plan and intent |
| | Suicidal Behaviour |
| CSSRS25 | Preparatory acts or behaviour |
| CSSRS23 | Aborted attempt |
| CSSRS21 | Interrupted attempt |
| CSSRS18 | Non-fatal suicide attempt |
| CSSRS27 | Completed suicide (only applicable for the post-baseline assessments) |
| | Self-Injurious Behaviour Without Suicidal Intent |
| CSSRS20 | Non-suicidal, self-injurious behaviour |

For patients with any post-baseline II/baseline III suicidal behaviour (C-SSRS scores of 6 to 10) or ideation (C-SSRS scores of 1-5), listings will be prepared including all C-SSRS scores; C-SSRS scores related to suicidal behaviour or ideation will be flagged.

## 12 Pharmacokinetic/Pharmacodynamic Analyses

Plasma concentrations of idalopirdine and memantine will be summarised descriptively for the APTS2 in the open-label treatment period with memantine.

## 13 Health Economic Analyses

The health economic assessments conducted during the open-label treatment period (RUD Lite, EQ-5D-3L and Dependence scale) in the open-label will be summarised by lead-in study. For the open label treatment period, absolute scores, change from Baseline I scores, and change from Baseline II will be summarised by visit week. The summaries of absolute scores and change from Baseline I scores will include data from the lead-in study and the open-label treatment period.

For the open label treatment period with memantine, absolute score and change from Baseline III in MMSE total score will be summarised by visit week.

## 14 Interim Analyses

No interim analyses planned.

 Trial Site Number: Study Level

LU Study Number: 14861B Pluto ID: CLI\_00933680 Status: Final


## 15 Sample Size Considerations

Open-label treatment period:

The study will include eligible patients who have completed Visit 7 (Completion Visit) of the lead-in studies. Assuming a completion rate of 85% and that approximately 85% of these are eligible and complete the extension study, this results in a total of approximately  $(3x310 + 3x280) \times 85\% \times 85\% \approx 1280$  patients completing this study.

*Open-label treatment period with memantine (sub-study):* 

With a sample size of n=100 the upper 1-sided 90% confidence limit for 0 to 10 AEs observed is:

| Number of AEs observed | 0 | 1 | 2 | 3 | 4 | 5 | 10 |
|---|---|---|---|---|---|---|---|
| Upper 1-sided CI for AE incidence | 2.3% | 3.9% | 5.3% | 6.6% | 7.9% | 9.1% | 15.0% |

This is regarded as sufficient accuracy for evaluating safety and tolerability.

## 16 Data and Analysis Standards and Statistical Software

The data will be collected and analysed in accordance with the Lundbeck standards specified in Lundbeck SDTM, Version 3.1.2 or later, SADs, Version 5.1 or later, and TGML, Version 7.0 or later.

The statistical software used will be SAS®, Version 9.4 or later.

## 17 Changes to Analyses Specified in the Protocol

C-SSRS will be summarized as worst case per treatment period rather than worst case per visit. However, all C-SSRS results for the study will be listed for those patients that experience any suicidal ideation or behaviour.

## 18 Details on Data Handling

#### 18.1 Definition of Baseline

The Baseline I value will be defined as the value captured either at the Screening Visit or the Baseline Visit of the lead-in study, whichever comes later.

Unless otherwise specified, the Baseline II Visit is the same as the Completion Visit (Visit 7/Week 24) in the lead-in studies (14861A and 14862A).

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Baseline III is the same as the Completion Visit (Visit 6/Week 28) of the open-label treatment period.

#### 18.2 Derived Variables

#### 18.2.1 MMSE Total Score and MMSE Stratum

MMSE consists of 8 subcategories (orientation to time, orientation to place, registration, attention and calculation, recall, language, repetition, and complex commands), with in total 30 questions recording correct/incorrect responses (coded 1/0). The MMSE total score is defined as the sum of the 30 questions and the total score ranges from 0 to 30 (at screening 12 to 22 due to inclusion criterion), with a lower scores meaning more severe dementia.

The subcategory *attention and calculation* consists of 5 questions (aCRF items MMSE04A to MMSE04E), where the patient continuously should subtract 7 from 100 (correct responses 93, 86, 79, 72, and 65). If a question is answered incorrectly and the subsequent questions not are recorded, the missing responses will be counted as incorrect (0).

The total score will be missing if three or more items scores are missing, and if less than three item scores are missing the missing item scores will be imputed by the worst case (0).

MMSE stratum (mild, MMSE total score ≥19; moderate, MMSE total score <19) used in the analyses will be based on the assessment collected at the lead-in study screening visit.

#### 18.2.2 ADAS-Cog Total Score

The ADAS-Cog assess the patient's orientation, memory (word recall, recognition, and remembering instructions), language (spoken language ability, comprehension of the spoken language, word finding difficulty, naming objects and fingers, following commands), and praxis (ideational and constructional). The ADAS-Cog total score is defined as the sum of the 11 item scores described in Panel 7. If three or more items scores are missing, the total score will be missing. If less than three item scores are missing item scores will be imputed by the worst score for the item.

The ADAS-Cog total score ranges from 0 to 70, with a lower score indicating a lower cognitive impairment.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Panel 7 Definition of ADAS-Cog Item Scores

| ADAS-Cog Item | Data collected in the eCRF (aCRF variable name) | Defintion of ADAS-Cog Item Scores used in the calculation of the total score (SADs paramed name) |
|---|---|---|
| 1. Word recall task | Total number of word recalled correctly, recorded in three trials (ranges 0-10 in each trial): ADCOG01 ADCOG02 ADCOG03 | Average of the total number of words recorded incorrectly in the three trials rounded to the closest integer with .5 rounded upwards (ranges from 0-10): ACITM01=round(((10- ADCOG01)+(10- ADCOG02)+(10- ADCOG03))/3,1.); If <3 of the eCRF scores are missing, the item score will be the average of the |
| 2. Naming task | Total number of object/fingers named <b>correctly</b> (ranges 0-17) ADCOG05 | available scores. eCRF score converted to total number of object/fingers named incorrectly (17-ADCOG05), and then classified according to the scoring scheme below (ranges 0-5): ACITM02= 0 = 0 - 2 1 = 3 - 5 2 = 6 - 8 3 = 9 - 11 4 = 12 - 14 5 = 15 - 17 |
| 3. Commands | Total number of commands performed <b>correctly</b> (ranges 0-5): ADCOG07 | eCRF score converted to total number of commands_performed incorrectly (ranges 0-5): ACITM03=5- ADCOG07; |
| 4. Constructional praxis | Total number of drawings performed <b>incorrectly</b> (ranges 0-5): ADCOG08 | ACITM04= ADCOG08 |
| 5. Ideational praxis | Total number of steps completed correctly (ranges 0-5): ADCOG09 | eCRF score converted to total number of steps completed incorrectly (ranges 0-5): ACITM05=5- ADCOG09; |
| 6. Orientation | Total number of items answered correctly (ranges 0-8): ADCOG10 | eCRF score converted to total number of items answered incorrectly (ranges 0-8): ACITM06=8- ADCOG10; |
| 7. Word recognition task | Total number of words identified <b>correctly</b> and total number of words identified <b>incorrectly</b> (both scores ranges 0-12): | Total number of words identified incorrectly, where scores>12 truncated to 12 (ranges 0-12): |

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final

Trial Site Number: Study Level


| | | A CITY 107 |
|---|---|---|
| | ADCOG11 | ACITM07= Min( (12, ADCOG11)+ ADCOG12, 12): |
| | ADCOG11 | Min( (12- ADCOG11)+ ADCOG12, 12); |
| | ADCOG12 | If ADCRGT01 or ADCRGT02 is missing, |
| | | the item score will be missing |
| 8. Remembering test instructions | Level of impairment (ranges 0-5, | ACITM08= ADCOG14 |
| 8 | see category labels below): | |
| | ADCOG14 | |
| | 0 = None | |
| | 1 = Very Mild<br>2 = Mild | |
| | 3 = Moderate | |
| | 4 = Moderately Severe | |
| | 5 = Severe | |
| 9. Language | Level of impairment (ranges 0-5, same category labels as for item 8): | ACITM09= ADCOG15 |
| | ADCOG15 | |
| 10. Comprehension of spoken language | Level of impairment (ranges 0-5, same category labels as for item 8): | ACITM10= ADCOG16 |
| | ADCOG16 | |
| 11. Word finding difficulty | Level of impairment (ranges 0-5, same category labels as for item 8): | ACITM11= ADCOG17 |
| | ADCOG17 | |

#### **18.2.3** ADCS-ADL<sub>23</sub> Total Score

The ADCS-ADL<sub>23</sub> scale contains of 23 item scores (See Panel 8), where each item contains one or more questions.

The ADCS-ADL<sub>23</sub> total score is defined as the sum of the 23 item scores. "Don't know" responses will be counted as worst case (0). For patients institutionalized, item score number 18 (Left On His/Her Own) will be counted as worst case (0). The scoring scheme for the item scores are described in Panel 8.

Trial Site Number: Study Level

LU Study Number: 14861B Pluto ID: CLI 00933680

Panel 8 ADCS-ADL<sub>23</sub> Items

| ADCS-ADL <sub>23</sub> Item | Data collected in the eCRF (aCRF variable name) | Defintion of ADCS-ADL <sub>23</sub> Item Scores used in the calculation of the total score (SADs paramed name) |
|---|---|---|
| 1. Usual Eating Performance | ADADL01 | Item score ranges 0-3: |
| | | ADL01=ADADL01 |
| 2. Optimal Walking<br>Performance | ADADL02 | Item score ranges 0-3: |
| 2 II 1 D 1/D1 11 | 1.0.1.0.1.0.2 | ADL02=ADADL02 |
| 3. Usual Bowel/Bladder Function | ADADL03 | Item score ranges 0-3: |
| | | ADL03=ADADL03 |
| 4. Usual Bathing Performance | ADADL04 | Item score ranges 0-3: |
| | | ADL04=ADADL04 |
| 5. Optimal Grooming<br>Performance | ADADL05 | Item score ranges 0-3: |
| | | ADL05=ADADL05 |
| 6. Dressing | ADADL06 | Item score ranges 0-7: |
| | ADADL07 | If ADADL06="No" or ADADL06="Don't know" then |
| | ADADL08 | ADL06=0; |
| | | else if ADADL06="Yes" then ADL06= |
| | | ADADL07; |
| 5 T | 1.0.1.0.0 | ADL06=ADL06+ADADL08; |
| 7. Use a Telephone | ADADL09 | Item score ranges 0-5: |
| | ADADL10 | If ADADL09="No" or |
| | | ADADL09="Don't know" then |
| | | ADL07=0;<br>else if ADADL09="Yes" then ADL07= |
| | | ADADL10; |
| 8. Watch Television | ADADL11 | Item score ranges 0-3: |
| | ADADL12 | if ADADL11="No" or |
| | A D A D L 12 | ADADL11="Don't know" then |
| | ADADL13 | ADL08=0;<br>%**"Yes"/"No"/"Don't know" counted |
| | ADADL14 | as 1/0/0; |
| | | else if ADADL11="Yes" then |
| | | ADL08= ADADL12+ADADL13+ |
| | | ADADL14; |

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final

Trial Site Number: Study Level


| 9. Pay Attention to Conversation | ADADL15 | Item score ranges 0-3: |
|---|---|---|
| | ADADL16 | If ADADL15="No" or ADADL15"Don't know" then ADL09=0; else if ADADL15="Yes" then ADL09= ADADL16; |
| 10. Clear Dishes | ADADL17 | Item score ranges 0-3: |
| | ADADL18 | If ADADL17="No" or<br>ADADL17="Don't know" then<br>ADL10=0;<br>else if ADADL17="Yes" then ADL10=<br>ADADL18; |
| 11. Find Belongings | ADADL19 | Item score ranges 0-3: |
| | ADADL20 | If ADADL19="No" or ADADL19="Don't know" then ADL11=0; else if ADADL19="Yes" then ADL11= ADADL20; |
| 12. Obtain Beverage | ADADL21 | Item score ranges 0-3: |
| | ADADL22 | If ADADL21="No" or ADADL21="Don't know" then ADL12=0; else if ADADL21="Yes" then ADL12= ADADL22; |
| 13. Make a Meal | ADADL23 | Item score ranges 0-4: |
| | ADADL24 | If ADADL23="No" or ADADL23="Don't know" then ADL13=0; else if ADADL23="Yes" then ADL13= ADADL24; |
| 14. Dispose of Garbage | ADADL25 | Item score ranges 0-3: |
| | ADADL26 | If ADADL25="No" or<br>ADADL25="Don't know" then<br>TADL14=0;<br>else if ADADL25="Yes" then ADL14=<br>ADADL26; |
| 15. Get Around Outside Home | ADADL27 | Item score ranges 0-4: |
| | ADADL28 | If ADADL27="No" or ADADL27="Don't know" then ADL15=0; else if ADADL27="Yes" then ADL15= ADADL28; |

Trial Site Number: Study Level

| 16.0.01 | 1 D 1 D1 20 | Tr. O.4 |
|---|---|---|
| 16. Go Shopping | ADADL29 | Item score ranges 0-4: |
| | ADADL30 | If ADADL29="No" or ADADL29="Don't know" then |
| | ADADL31 | ADL16=0;<br>%**"Yes"/"No"/"Don't know" counted |
| | | as 1/0/0 (ADADL31); |
| | | else if ADADL29="Yes" then<br>ADL16= ADADL30+ ADADL31; |
| 17. Keep Appointments | ADADL32 | Item score ranges 0-3: |
| 17. Heep rippointments | | |
| | ADADL33 | If ADADL32="No" or<br>ADADL32="Don't know" then |
| | | ADL17=0; |
| | | else if ADADL32="Yes" then ADL17= |
| 18. Left On His/Her Own | ADADL34 | ADADL33; |
| 18. Left On His/Her Own | ADADL34 | Item score ranges 0-3: |
| | ADADL35 | If ADADL34="Checked" then ADL18=0; |
| | ADADL36 | else if ADADL35="No" or<br>ADADL35="Don't know" then |
| | | ADL18=0; |
| | ADADL37 | %**"Yes"/"No"/"Don't know" counted |
| | ADADL38 | as 1/0/0;<br>else if ADADL35="Yes" then |
| | | ADL18= ADADL36+ ADADL37+ |
| 10 77 11 11 17 77 | 1.5.15.40 | ADADL38; |
| 19. Talk About Current Events | ADADL39 | Item score ranges 0-3: |
| | ADADL40 | if ADADL39="No" or |
| | ADADL41 | ADADL39="Don't know" then ADL19=0; |
| | TIDINDE TI | %**"Yes"/"No"/"Don't know" counted |
| | ADADL42 | as 1/0/0; |
| | | else if ADADL39="Yes" then<br>ADL19= ADADL40+ ADADL41+ |
| | | ADADL42; |
| 20. Read More Than 5 Minutes | ADADL43 | Item score ranges 0-2: |
| | ADADL44 | if ADADL43="No" or |
| | ADADL45 | ADADL43="Don't know" then ADL20=0; |
| | ADADL <del>I</del> J | %**"Yes"/"No"/"Don't know" counted |
| | | as 1/0/0; |
| | | else if ADADL43="Yes" then<br>ADL20= ADADL44+ ADADL45; |
| 21. Write Things Down | ADADL46 | Item score ranges 0-3: |
| | ADADL47 | If ADADL46="No" or |
| | | ADADL46="Don't know" then |
| | | ADL21=0;<br>else if ADADL46="Yes" then ADL21= |
| | | ADADL47; |
| | l | , |

| 22. Perform Pastime | ADADL48 | Item score ranges 0-3: |
|---|---|---|
| | ADADL49 | If ADADL48="No" or<br>ADADL48="Don't know" then<br>ADL22=0;<br>else if ADADL48="Yes" then ADL22=<br>ADADL49; |
| 23. Use Household Appliance | ADADL50 | Item score ranges 0-4: |
| | ADADL51 | If ADADL50="No" or<br>ADADL50="Don't know" then<br>ADL23=0;<br>else if ADADL50="Yes" then ADL23=<br>ADADL51; |

If five or more items scores are missing, the total score will be missing. If less than five item scores are missing, the missing questions within the item score will be imputed by the worst case for each missing question (missing main responses will be imputed by 0; if the main response equal to "Yes", missing subsequent question(s) will be imputed by the worst score for each question).

The ADCS-ADL<sub>23</sub> total score ranges from 0 to 78, with a higher score indicating a higher functioning status.

#### 18.2.4 NPI Total Score and Individual Items

The NPI scale consists of 12 domains (Delutions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, Aberrant Motor Behaviour, Sleep, and Appetite and Eating Disorders). The NPI total score is defined as the sum of the 12 domain scores, where the domain score for each domain is calculated as (the domain is given by category 1-12 in the aCRF variable NPI01):

- If status (aCRF NPI02) is equal to "Not Applicable" or "No", the NPI domain score will be equal to 0; otherwise, the NPI domain score will be the product of frequency (aCRF NPI03, ranging from 1 to 4), and severity (aCRF NPI04, ranging from 1 to 3).
- If four or more domain scores are missing (due to missing record in status, or missing frequency, or severity for the domain), the NPI total score will be missing. If less than four domain scores are missing, the missing doimains will in the calculation of the NPI total score be imputed by the mean of the non-missing domain scores, rounded to the closest integer (.5 rounded upwards).

Each domain score ranges from 0 to 12, and the NPI total score ranges from 0 to 144 with a higher score indicates a more serious behavioral issue.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680


#### 18.3 **Assigning Data to Visits**

#### 18.3.1 **Rating Scales**

The assessment at the Withdrawal Visit for patients withdrawn from treatment will be assigned to a nominal visit in the Treatment Period, according to the visit windowing specified in Panel 9 and Panel 10. The assessment collected at the scheduled visit will be used in the analyses, or the windowed assessment from the Withdrawal Visit if no schedule assessment is available. If the assessment at the Withdrawal Visit is assigned to the same visit as an assessment at a scheduled visit, the assessment from the scheduled visit will be used. Otherwise, the assessments at the scheduled visits will be used.

Panel 9 **Visit Windows for Efficacy Assessments (open-label treatment period)** 

| Nominal Visit Number | Nominal Visit Week | Nominal Visit Day | Time Window |
|---|---|---|---|
| V1 (Baseline II /Completion Visit for lead-in study) | 0 | 0 | 0 |
| V4 | 12 | 84 | 1 to 139 |
| V6 (Completion/Withdrawal) | 28 | 196 | >139 |

MMSE is only assessed at Baseline II, Baseline III and the Completion/Withdrawal visit. As such, the visit windows for MMSE are specified in Panel 10.

Panel 10 Visit Windows for MMSE

| Nominal Visit Number | Nominal Visit Week | Nominal Visit Day | Time Window |
|---|---|---|---|
| V1 (Baseline II /Completion Visit for leadin study) | 0 | 0 | 0 |
| V6 (Baseline III/Completion Visit for open-<br>label treatment period) | 28 | 196 | 1 to 279 |
| V11 (Completion Visit for open-label treatment period with memantine) | 52 | 364 | >279 |

#### 18.3.2 Safety Variables

The first usable assessment at the Withdrawal Visit for safety variables (laboratory tests, vital signs, weight and ECGs) will be assigned to a nominal visit in the corresponding Treatment Period, according to the visit windowing specified in Panel 11.

For assessments at the Baseline II/III Visit, the last usable assessment will be used. For assessments at visits post-baseline, the first usable assessment from the scheduled visit will be used, or the assessment from the Withdrawal Visit will be used if no scheduled assessment is available.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Panel 11 Visit Windows for Safety Assessments

| Nominal Visit Number | Nominal Visit<br>Week | Nominal Visit Day | Time Window |
|---|---|---|---|
| Open-label treatment period | | | |
| V1 (Baseline II/Completion Visit for lead-in study) | 0 | 0 | 0 |
| V2 | 4 | 28 | 1 to 41 |
| V3 | 8 | 56 | 42 to 69 |
| V4 | 12 | 84 | 70 to 111 |
| V5 | 20 | 140 | 112 to 167 |
| V6 (Completion Visit for open-label treatment period) | 28 | 196 | >167 |
| Open-label treatment period with memantine (APTS2) | | | |
| V6 (Baseline III/Completion Visit open-label treatment period) | 28 | 196 | 167 to 209 |
| V8 | 32 | 224 | 210 to 237 |
| V9 | 36 | 252 | 238 to 265 |
| V10 | 40 | 280 | 266 to 321 |
| V11 (Completion visit for open-label treatment period with memantine) | 52 | 364 | >321 |

#### 18.4 Handling of Missing or Incomplete Dates/Times

#### **18.4.1 IMP Start and Stop Dates**

A missing IMP start date will be imputed with the date of Baseline II for patients in the APTS with an unknown IMP start date.

A missing IMP stop date will not be imputed. As such, exposure will be missing for a patient with a missing IMP stop date and the patient will contribute as having no exposure in the calculation of PYE. If it can be ascertained from other data that the patient did take IMP until a specific date, this date may be used to calculate exposure.

#### 18.4.2 Withdrawal Date

For withdrawn patients with a missing Withdrawal Visit, the date of the last attended visit in the corresponding Treatment Period will be used in the calculation of time to withdrawal from treatment.

#### 18.4.3 Medical Disorder Start and Stop Dates

No imputation of dates will be done.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

#### **18.4.4** Adverse Event Start and Stop Dates

If a stop date is missing due to an adverse event being on-going, the last visit date will be used as the stop date in the classification of TEAEs.

An adverse event with a missing or incomplete start or stop date will be classified as a pretreatment adverse event if the patient was taking placebo in the lead-in study and the following conditions are met:

- The start date is missing or incomplete, and the stop date is prior to the Baseline II visit, or the stop date is incomplete but known to be prior to the Baseline II visit (stop day is missing and stop year and month are before the year and month of the Baseline II visit, or stop day and month are missing and stop year is before the year of Baseline II)
- The start date is incomplete but known to be prior to the Baseline II visit (start day is missing and start year and month are before the year and month of the Baseline II visit, or start day and month are missing and start year is before the year of the Baseline II visit), and no change in intensity

If a start date is missing for an adverse event and the stop date is prior to the Baseline II visit, then the adverse event will be regarded as starting prior to the study and will not be included in the reporting of AEs in the study. In all other instances of an adverse event with a missing start or stop date, the adverse event will be classified as a TEAE.

#### **18.5** Grouping of Small Countries

In analyses where country is a factor, countries where not all treatment groups are represented in the APTS will be grouped according to the following stepwise procedure:

- Step 1 All countries where not all treatment groups are represented in the APTS will be grouped into a single collective country within the same continent.
- Step 2 If not all treatment groups are represented in the APTS for a grouped country, the countries will be grouped with the smallest country within the same continent for which all treatment groups are represented in the APTS. If there is more than one such country, the first country in ascending alphabetic order will be selected for the grouping.

Version: 10

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

Status: Final
### References

1. United States Food and Drug Administration (FDA). Guidance for Industry: Drug-induced liver injury: Premarketing Clinical Evaluation. July 2009.

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

# Appendix I Statistical Analysis Plan Authentication and Authorisation

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final

Trial Site Number: Study Level


## Statistical Analysis Plan Authentication and Authorisation

| Study title: | An open-label extension study to evaluate the long-term safety and tolerability of Lu AE58054 as adjunctive treatment to donepezil in patients with mild-moderate Alzheimer's disease |
|---|---|
| SAP date: | 10 July 2017 |
| This document has been sign | ed electronically. The signatories are listed below. |
| Authentication | |
| Biostatistician: | |
| CRS: | , CRD Neurology Idalopirdine Team |
| Authorisation | |
| Head of Biostatistics: | |

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI\_00933680

Pluto ID: CLI\_00933680 Status: Final Version: 1.0

# Appendix II Study Flow Chart

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI\_00933680

# **Study Flow Chart**

#### Study Procedures and Assessments [open-label treatment period]

| Visit | Baseline<br>II <sup>a</sup> | , | Treatme | nt Perio | d | Completion/<br>Withdrawal <sup>b</sup> | Safety Follow-up <sup>c</sup> |
|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Day <sup>d</sup> / | 0 | 28/ | 56/ | 84/ | 140/ | 196/ | 224/ |
| End of Week | | 4 | 8 | 12 | 20 | 28 | 32 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ± 7d | ± 7d | ± 7d | ± 7d | ± 7d | + 7d |
| Screening/Baseline Proced | ures and As | ssessmer | nts | | | | |
| Signed informed consent | √ | | | | | | |
| Demographics | $\sqrt{f}$ | | | | | | |
| Height | $\sqrt{f}$ | | | | | | |
| Medical history | $\sqrt{f}$ | | | | | | |
| Inclusion/exclusion criteria | $\sqrt{}$ | | | | | | |
| Efficacy Assessments | | | * | * | | | |
| MMSE | √g | | | | | <del>-</del> | |
| ADAS-Cog | √g | | | $\sqrt{}$ | | √ | |
| ADCS-ADL <sub>23</sub> | √g | | | | | $\sqrt{}$ | |
| ADCS-CGIC <sup>h</sup> | √g | | | $\checkmark$ | | $\sqrt{}$ | |
| NPI | $\sqrt{g}$ | | | $\sqrt{}$ | | $\sqrt{}$ | |
| Other Assessments | | | | | | | |
| RUD Lite | √g | | | √ | | √ | |
| EQ-5D-3L | $\sqrt{g}$ | | | $\checkmark$ | | $\sqrt{}$ | |
| Dependence scale | $\sqrt{i}$ | | | $\checkmark$ | | $\sqrt{}$ | |
| Safety Assessments | | | | | | | |
| Adverse events | $\sqrt{j}$ | | √ | √ | √ | √ | $\sqrt{k}$ |
| Blood and urine sampling | | | | | | | |
| for clinical safety | lσ | 1 | 1 | 1 | 1 | 1 | |
| laboratory tests | √g<br>. /g | <b>V</b> | <b>V</b> | <b>V</b> | N<br>I | V | |
| Vital signs, weight, ECGs<br>C-SSRS | √g<br>√g | <b>V</b> | <b>\</b><br>! | <b>V</b> | <b>N</b><br>l | <b>V</b> | |
| Examinations (physical, | .γ° | ٧ | ٧ | ٧ | ٧ | V | |
| neurological) | √g | | √ | | √ | √ | |
| Other Study Procedures | | | | | | | |
| IMP and donepezil <sup>1</sup> | -1 | . 1 | .1 | .1 | ا ۽ | | |
| hydrochloride dispensed | V | <b>V</b> | √<br>! | <b>V</b> | N | 1 | |
| IMP and donepezil <sup>l</sup> | | ٧ | V | V | V | V | |


LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final


| Visit | Baseline<br>II <sup>a</sup> | r | Гreatme | nt Perio | d | Completion/<br>Withdrawal <sup>b</sup> | Safety Follow-up |
|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Day <sup>d</sup> / | 0 | 28/ | 56/ | 84/ | 140/ | 196/ | 224/ |
| End of Week | | 4 | 8 | 12 | 20 | 28 | 32 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ± 7d | ± 7d | ± 7d | ± 7d | ± 7d | + 7d |
| Screening/Baseline Proced | lures and As | ssessmer | its | | | | |
| hydrochloride returned accountability tracked | | | | | | | |
| Recent and concomitant medication | √j | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\checkmark$ |
| Dispense Patient<br>Identification card | $\sqrt{}$ | | | | | | |
| Patient Identification card returned | | | | | | $\sqrt{m}$ | |
| Informed Consent<br>Provided<br>[open-label treatment<br>period with memantine | | | | | | | |
| period with memantine | | | | | ln | | |

- a. For the purposes of clarity, the Baseline Visit is called Baseline II Visit and this visit is the same as Visit 7 (Completion Visit) in the lead-in study.
- b. This visit should take place as soon as possible after the patient withdraws from the study.
- c. Patients who complete the study and do not enter into the open-label treatment period with memantine (sub-study) will have a Safety Follow-up Visit which is at least 4 weeks (+ up to 7 days) after the last dose of IMP. Patients withdrawn will likewise be followed-up 4 weeks (+ up to 7 days) after withdrawal except for those who withdraw their consent. Patients who withdraw their consent should still have a safety follow-up, but the visit must only be recorded in the medical records.
- d. All assessments can be completed over a maximum of two consecutive days, in this case the first day should be considered as the visit day of the study. Note: If a visit takes place over two consecutive days the IMP should be dispensed on the second day, after all assessments have been performed. For visits other than the Baseline II visit, the visit window must allow for the previously dispensed IMP to last for both visit days.
- e. If the date of a patient visit does not conform to the study plan, subsequent visits should be planned to maintain the visit schedule relative to Baseline II. Number of days between 2 visits must not exceed the number of days for which IMP is provided in the wallet cards.
- f. Lead-in study screening visit (Visit 1) data transferred.
- g. Assessments and procedures conducted at Visit 7 (Completion Visit) of the lead-in study will be transferred and will not be repeated at the Baseline II Visit of this extension study.
- h. During evaluation the patient should be compared to Baseline I assessment of the lead-in study.
- i. Data will be transferred from Visit 7 (Completion Visit) of the lead-in study or entered manually to the eCRF if the scale has been administered for the first time at Visit 1 of the extension study.
- j. On-going adverse events and Concomitant Medications at Visit 7 (Completion Visit) from the lead-in study are to be transferred to the eCRF.
- k. Only for adverse events on-going at Completion/Withdrawal Visit and new SAEs.
- 1. As base treatment, donepezil hydrochloride 10 mg/day will be dispensed as wallet cards.
- m. *Patient Identification Card* should only be returned after the last dose of IMP has been taken, that is at the end of the treatment period.

(substudy)]

n. For patients who may be eligible to participate in the open-label treatment period with memantine (substudy), it is suggested that the *Informed Consent Form* is provided.

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final


#### Study Procedures and Assessments [open-label treatment with memantine (sub-study)]

| Visit | Baseline<br>III <sup>a</sup> Treatment Period | | | | Completion/ Safety<br>Withdrawal <sup>b</sup> Follow-up <sup>c</sup> | |
|---|---|---|---|---|---|---|
| Visit Number | 6 | <b>8</b> <sup>j</sup> | 9 | 10 | 11 | 12 |
| Day/ <sup>d</sup> | 0 | 224/ | 252/ | 280/ | 364/ | 392/ |
| End of Week | | 32 | 36 | 40 | 52 | 56 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ± 7d | ±7d | ± 7d | ±7d | + 7d |
| Screening/Baseline Procedures and Assessments | | | | | | |
| Signed informed consent | | | | | | |
| Demographics, height | $\sqrt{}$ | | | | | |
| Medical history | $\sqrt{}$ | | | | | |
| Inclusion/exclusion criteria | $\sqrt{}$ | | | | | |
| Efficacy Assessments | | | | | | |
| MMSE | √ f | | | | √ | |
| Pharmacoeconomic Assessments | | | | | | |
| Patient's current living accommodation (question extracted from the RUD-Lite) | √ f | | | $\sqrt{}$ | V | |
| Dependence scale | $\sqrt{f}$ | | | $\sqrt{}$ | $\checkmark$ | |
| Pharmacokinetic Assessments | | | | | | |
| Blood sampling for idalopirdine and memantine | √ | √ | √ | | √ | |
| Safety Assessments | | | | | | |
| Adverse events | $\sqrt{f}$ | √ | √ | | √ | $\sqrt{\mathrm{g}}$ |
| Blood and urine sampling for clinical safety laboratory tests | $\sqrt{\mathrm{f}}$ | $\sqrt{}$ | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | |
| Vital signs, weight, ECGs | $\sqrt{f}$ | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | $\sqrt{}$ | |
| C-SSRS | $\sqrt{f}$ | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | $\sqrt{}$ | |
| Examinations (physical, neurological) <b>Other Study Procedures</b> | √ <sup>f</sup> | | | √<br>√ | √ | |
| IMP and donepezil hydrochloride dispensed. Memantine prescribed h | √ | √ | √ | | | <del></del> |
| IMP, memantine and donepezil hydrochloride returned and accountability tracked h | | $\checkmark$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | |
| Recent and concomitant medication | $\sqrt{\mathrm{f}}$ | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | $\checkmark$ | |
| Dispense Patient Identification card | $\sqrt{}$ | | | | | |
| Patient Identification card returned | | | | $\sqrt{i}$ | | |

LU Study Number: 14861B Pluto ID: CLI\_00933680 Status: Final

Trial Site Number: Study Level


- a. The Baseline Visit for this study (Baseline III) is the same visit as Visit 6 (end of Week 28) for patients who complete the open-label treatment period.
- b. This visit should take place as soon as possible after the patient withdraws from the study.
- c. Patients who complete the study will have a Safety Follow-up Visit which is at least 4 weeks (+ up to 7 days) after the last dose of IMP. Patients withdrawn will likewise be followed-up 4 weeks (+ up to 7 days) after withdrawal except for those who withdraw their consent. Patients who withdraw their consent should still have a safety follow-up, but the visit must only be recorded in the medical records.
- d. All assessments can be completed over a maximum of two consecutive days, in this case the first day should be considered as the visit day of the study. Note: If a visit takes place over two consecutive days the IMP should be dispensed on the second day, after all assessments have been performed. For visits other than the Baseline Visit of this study, the visit window must allow for the previously dispensed IMP to last for both visit days.
- e. If the date of a patient visit does not conform to the study plan, subsequent visits should be planned to maintain the visit schedule relative to Baseline III of this study. Number of days between 2 visits must not exceed the number of days for which IMP is provided in the wallet cards.
- f. Assessments and procedures are the same as Visit 6 in the open-label treatment period.
- g. Only for adverse events on-going at Completion/Withdrawal of this study and new SAEs.
- h. Donepezil hydrochloride 10 mg/day will be dispensed as wallet cards. Memantine (titration doses plus patient's individualised maintenance dose) will be prescribed by the investigator or another medically-qualified person and the investigator should make sure that an adequate supply of memantine is prescribed to last between two visits (including visit windows). In addition to the return of IMP and donepezil hydrochloride, patient will be asked to bring used and unused memantine in original packaging to the visit for accountability purposes.
- i. *Patient Identification Card* should only be returned after the last dose of IMP has been taken, that is at the end of the treatment period.
- j. All patients entering the open-label treatment period with memantine (sub-study) will perform Visit 8 right after Visit 6 [Visit 7 is the Safety Follow-up visit only for patients who do not continue into the open-label treatment period with memantine (sub-study)].

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI 00933680

# Appendix III SAS® Code

LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final Version: 1.0

### SAS® Code

```
The SAS code for the MMRM-analysis (for each lead-in study) will be:

%**MMSTR=MMSE stratum;

proc mixed noclprint data=ADAS ic method=REML;

class usubjid country analysis_week armcd MMSSTR;

model ADASTOT_DL = ADASTOT_BL MMSSTR country armcd analysis_week

armcd*analysis_week MMSSTR*analysis_week ADASTOT_BL*analysis_week

/s DDFM=KR;

repeated analysis_week/subject=usubjid type=un;

run;
```

 LU Study Number: 14861B Trial Site Number: Study Level

Status: Final Version: 1.0

Pluto ID: CLI 00933680

# Appendix IV PCS Criteria

LU Study Number: 14861B Trial Site Number: Study Level Pluto ID: CLI\_00933680

### **PCS** Criteria

Table 1 PCS Criteria for Clinical Safety Laboratory Tests

| CDISC term | Test (units) | PCS Low | PCS High |
|---|---|---|---|
| Liver | | | |
| AST | S-aspartate aminotransferase (IU/L) | | $\geq 3 \times ULN$ |
| ALT | S-alanine aminotransferase (IU/L) | | $\geq$ 3 × ULN |
| BILI | S-bilirubin (μmol/L) | | ≥ 34 |
| BILDIR | S-direct bilirubin (µmol/L) | | ≥ 12 |
| ALP | S-alkaline phosphatase (IU/L) | | $\geq 3 \times ULN$ |
| GGT | S-gamma glutamyl transferase (IU/L) | | $\geq 200$ |
| Kidney | | | |
| CREAT | S-creatinine (µmol/L) | | $\geq 1.5 \times ULN$ |
| BUN | B-urea nitrogen (mmol/L) | | ≥ 11 |
| Electrolytes | | | |
| SODIUM | S-sodium (mmol/L) | ≤ 125 | ≥ 155 |
| K | S-potassium (mmol/L) | ≤ 3.0 | $\geq 6.0$ |
| CA | S-calcium (mmol/L) | ≤ 1.8 | $\geq 3.0$ |
| BICARB | S-bicarbonate (mmol/L) | ≤ 12 | ≥ 38 |
| Endocrine/Meta | bolic | | |
| GLUC | Serum glucose (mmol/L) | ≤ 3.9 | ≥ 11.1 |
| GLUC | Serum glucose, fasting (mmol/L) | ≤ 3.5 | $\geq 7.0$ |
| TSH | S-thyrotropin (mIU/L) | ≤ 0.3 | ≥ 5.5 |
| ALB | Albumin (g/L) | ≤ 27 | |
| Lipids | | | |
| CHOL | S-cholesterol (mmol/L) | | ≥ 7.8 |
| CHOL | S-Cholesterol, fasting (mmol/L) | | $\geq 6.2$ |
| TRIG | Triglycerides (mmol/L) | | ≥ 5.65 |
| TRIG | Triglycerides, fasting (mmol/L) | | ≥ 4.2 |
| Haematology/Co | pagulation | | |
| INR | P-INR (Prothrombin ratio) | | $\geq 2.0$ |
| PLAT | B-thrombocytes platelet count (×10E9/L) | ≤ 75 | $\geq 600$ |
| HGB | B-haemoglobin (g/dL) | ≤ 9.5 (women)<br>≤ 11.5 (men) | ≥ 16.5 (women)<br>≥ 18.5 (men) |
| RBC | B-erythrocytes (×10E12/L) | ≤ 3.5 (women)<br>≤ 3.8 (men) | $\geq$ 6.0 (women)<br>$\geq$ 7.0 (men) |
| WBC | B-Leukocytes (×10E9/L) | $\leq$ 2.8 | ≥ 16 |
| NEUTLE | B-Neutrophils/leukocytes (%) | $\leq 20$ | ≥ 85 |
| EOSLE | B-eosinophils/leukocytes (%) | | ≥ 10 |


LU Study Number: 14861B Pluto ID: CLI\_00933680

Status: Final


| CDISC term | Test (units) | PCS Low | PCS High |
|------------|------------------------------|---------|------------|
| BASOLE | B-basophils/leukocytes (%) | | ≥ 10 |
| LYMLE | B-Lymphocytes/leukocytes (%) | ≤ 10 | ≥ 75 |
| MONOLE | B-Monocytes /leukocytes (%) | | ≥ 15 |
| Infection | | | |
| CRP | S-C-reactive protein (mg/L) | | ≥ 25 |
| Urine | | | |
| GLUC | U-Glucose | | Increase≥2 |
| KETONES | U-Ketones | | Increase≥2 |
| OCCBLD | U-Occult Blood | | Increase≥2 |

Table 2 PCS Criteria for Vital Signs and Weight

| CDISC term | Variable (units) | <b>PCS Criterion Low</b> | PCS Criterion High |
|---|---|---|---|
| WEIGHT | Weight (kg) | Decrease ≥ 7% | Increase ≥ 7% |
| BMI | Body mass index (kg/m2) | Decrease $\geq 7\%$ | Increase $\geq 7\%$ |
| DIABP | Supine diastolic blood pressure (mmHg) | $\leq$ 50 and decrease $\geq$ 15 | $\geq 105$ and increase $\geq 15$ |
| SYSBP | Supine systolic blood pressure (mmHg) | $\leq$ 90 and decrease $\geq$ 20 | $\geq 180$ and increase $\geq 20$ |
| PULSE | Pulse rate supine/sitting/unknown (bpm) | $\leq$ 50 and decrease $\geq$ 15 | $\geq$ 120 and increase $\geq$ 15 |

**Table 3** PCS Criteria for ECG Parameters

| CDISC term | Parameter (units) | <b>PCS Criterion Low</b> | <b>PCS Criterion High</b> |
|---|---|---|---|
| <b>Absolute Time Int</b> | erval | | |
| PRMEAN | PR interval (msec) | | ≥ 260 |
| QRSDUR | QRS interval (msec) | | ≥ 150 |
| QTMEAN | QT interval (msec) | | ≥ 500 |
| <b>Derived Time Inte</b> | rval | | |
| QTcB | QTcB interval (msec) | < 300 | > 500 or increase > 60 |
| QTcF | QTcF interval (msec) | < 300 | > 500 or increase > 60 |
| HRMEAN | ECG Mean heart rate (beats/min) | $\leq$ 50 and decrease $\geq$ 15 | $\geq$ 120 and increase $\geq$ 15 |

Trial Site Number: Study Level
